CLINICAL TRIAL: NCT06674746
Title: The Effect of Solution-Focused Approach on the Internet, Social Media Addiction and Self-Efficacy Levels of Nursing Students
Brief Title: Effect of Solution-Focused Approach on the Internet,Social Media Addiction and Self-Efficacy Levels OfNursing Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Taha Yasir Mert, Principal Investigator, Cumhuriyet University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 17082022
Record Dates: First submitted 2022-09-16; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Risk Behavior; Social Media Addiction; Internet Addiction
Keywords: solution focused approach; nursing; internet addiction; social media addiction; self-efficacy-sufficiency
MeSH Terms: conditions — Risk-Taking; Internet Addiction Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Using the simple random numbers table from the population in the risk group, 60 randomly selected students will be randomly assigned to the experimental and control groups as 30 students. A two-stage stratified random method will be used in order to make assignments to the intervention and control groups equally and homogeneously. Firstly; The class and gender strata determined by scanning the literature will be created. Afterwards, each class and the male and female students in these classes will be determined. Then, the students in each stratum will be assigned to the intervention and control groups according to the two-layer random method, one intervention and one control.
  Interventions: Behavioral: SOLUTION FOCUSED APPROACH
- control (No Intervention): Using the simple random numbers table from the population in the risk group, 60 randomly selected students will be randomly assigned to the experimental and control groups as 30 students. A two-stage stratified random method will be used in order to make assignments to the intervention and control groups equally and homogeneously. Firstly; The class and gender strata determined by scanning the literature will be created. Afterwards, each class and the male and female students in these classes will be determined. Then, the students in each stratum will be assigned to the intervention and control groups according to the two-layer random method, one intervention and one control.

INTERVENTIONS:
Behavioral: SOLUTION FOCUSED APPROACH — The interviews with the control group were planned as eight sessions. There will be defined time intervals between sessions. It is estimated to take 6 months.
  Arms: intervention

SUMMARY:
The purpose of this research; is to determine the effect of solution-oriented approach on internet, social media addiction and self-efficacy levels of nursing students.

A pretest-posttest randomized controlled experimental design will be used in the research.

DETAILED DESCRIPTION:
The research will be carried out between 4 April 2022 and 28 April 2023 at Sivas Cumhuriyet University . Personal Information Form, Internet Addiction Scale, Social Media Addiction Scale and Self-Efficacy Competence Scale were applied to a total of 1057 nursing students who were continuing their education in the 1st, 2nd and 3rd years at the Faculty of Health Sciences (683) and Suşehri Health College (374), where the research would be conducted.Since the final data of the study will be received next year, students in the 1st, 2nd and 3rd grades will be included in the interviews in order to prevent data loss, and 4th graders will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25,
* 67 < Internet Addiction Scale (IAS) Score < 109,
* 73 < Social Media Addiction (SMDS) Score < 140.

Exclusion Criteria:

* Receiving any psychological counseling and treatment,
* Being closed to communication,
* To have extended the term,
* Not volunteering to participate in the research.

Ages: 18 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-10-24 (Actual); Study Completion 2023-10-24 (Actual)

PRIMARY OUTCOMES:
Internet Addiction Scale | 10 minute
  Developed by Günç and Kayri (2010), the İBÖ is in the five-point likert type, and the likert-style expressions are; "Strongly Agree", "Agree", "Undecided", "Disagree", "Strongly Disagree".
Social Media Addiction Scale | 10 minute
  The Social Media Addiction Scale was developed by Tutgun-Ünal and Deniz (2015) in order to measure the social media addiction of university students and all validity and reliability studies were carried out. Consisting of 41 items and four factors (occupation, mood regulation, repetition, and conflict), SMDS is a 5-point Likert-type scale graded as "Always", "Often", "Sometimes", "Rarely" and "Never".
Self-Efficacy-Efficacy Scale | 5 minute
  The Self-Efficacy Efficiency scale, developed by Sherer et al. (1982) and adapted into Turkish by Gözüm and Aksayan (1999), is a 5-point Likert-type scale and includes 23 items. The cronbach alpha internal consistency coefficient of the Turkish version of the scale was found to be .81 (Gözüm & Aksayan, 2010).

CONTACTS AND LOCATIONS:
Overall Officials: Taha Mert, postgraduate, Study Director — Cumhuriyet University; Nuran Güler, professor, Study Director — Cumhuriyet University